CLINICAL TRIAL: NCT06368089
Title: Short Effects of Speci|c Inspiratory Muscle Training and Early Mobilization in Prolonged Mechanically Ventilated Patients
Brief Title: Short Effects of SIMT and EM in Prolonged Mechanically Ventilated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Saikaew Chuachan, Department of Physical Therapy, Faculty of Medicine, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC.66-474-30-2; MR-PSU:66-30-21-406 (Other Grant/Funding Number: Faculty of Medicine, Prince of Songkla University)
Record Dates: First submitted 2024-04-01; First posted 2024-04-16 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Ventilator Dependent
Keywords: Specific inspiratory muscle training; Early mobilization; Lung compliance; Prolong mechanical ventilation; Weaning outcome
MeSH Terms: interventions — Population Groups; Early Ambulation

STUDY DESIGN:
Intervention Model Description: randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT group (Experimental): Inspiratory muscle training group
  Interventions: Other: Inspiratory muscle training (IMT) group
- EM group (Active Comparator): Early mobilization group
  Interventions: Other: Early mobilization (EM) group

INTERVENTIONS:
Other: Inspiratory muscle training (IMT) group — The IMT group receives inspiratory muscle training of 50%MIP, 6 breaths/set 10 sets/day for 7 days combined with conventional chest physiotherapy including; percussion, vibration, postural draining, positioning, and passive range of motion.
  Arms: IMT group
Other: Early mobilization (EM) group — The ER group received active exercise in sitting, standing, and marching 30 minutes/day for 7 days with conventional chest physical therapy
  Arms: EM group

SUMMARY:
Using mechanical ventilation for more than 18 hours can affect respiratory muscle and postural muscle control, making it difficult to wean off the ventilator and reducing mobility. The aim of this study is to:

1. Compare the effects of respiratory muscle strength training and early mobilization on dynamic lung compliance and maximum inspiratory pressure before and after a 7-day training period.
2. Compare the success rate of weaning and the duration of weaning between the respiratory muscle strength training and the early mobilization program.

DETAILED DESCRIPTION:
The prolonged mechanical ventilation results in difficulty weaning off the ventilator. Inspiratory muscle strength and early mobilization can contribute to the expansion of lung parenchyma and facilitate success in weaning off respiratory support. Thus, this study aimed to explain the impact of inspiratory muscle training and early mobilization on dynamic lung compliance, spontaneous breathing time, and success rate in patients who have undergone mechanical ventilation for more than 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patients with respiratory diseases who have been on mechanical ventilation for more than 48 hours and are ready to be weaned off or undergoing weaning trials with continuous positive airway pressure (CPAP) or synchronized intermittent mandatory ventilation (SIMV).
* The PaO2/FiO2 ratio is ≥ 150-200, with FiO2 ≤ 0.4-0.5 and PEEP ≤ 5-8 cmH2O, and a pH > 7.3 in blood plasma.
* The age range is between 40 and 80 years old.
* Patients exhibit good self-awareness and cooperation in training (Riker score of 4).
* They can understand and communicate in Thai

Exclusion Criteria:

* Clinical instability (HR > 120 beats/minute, RR > 30 breaths/minute, SatO2 < 90%, SBP > 140 mmHg or < 90 mmHg)
* Patients who can be extubated and use non-invasive ventilation only or successfully extubated within the first 24 hours.
* Patients with altered mental status (Glasgow Coma Score < 10) and inability to cooperate with training (Riker score < 4 or > 4)
* Patients with limitations or contraindications such as inability to adjust the bed to a 45-degree angle or sit on the side of the bed, such as those with spinal cord injuries or recent head surgeries.
* History of hemoptysis, pneumothorax
* History of neuromuscular diseases causing muscle weakness and decreased sensation.
* Patients with excessive cardiac stimulation (> 5 micrograms per kilogram per minute)
* Heart rate > 140 beats per minute
* Hemoglobin levels < 8-10 grams per deciliter
* Patients with difficult airway issues.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Maximum inspiratory pressure (MIP) | baseline and day 7 after program
  MIP measurement using manometer, the device can be attached directly to the ETT or tracheostomy tube, and measures the pressure generated by patient on inhalation against a closed system.
Dynamic lung compliance (Cdyn) | baseline and day 7 after program
  Dynamic lung compliance refers to the ratio of the change in volume to the change in pressure over a tidal breath, with the pressure measured at moments of zero flow during breathing that recording from the mechanical ventilation

SECONDARY OUTCOMES:
Weaning time | baseline and day 7 after program
  Duration of weaning time (hour)
Weaning outcome | baseline and day 7 after program
  measure weaning success rate
Grip strength | baseline and day 7 after program
  using hand grip dynamometer
chest wall expansion | baseline and day 7 after program
  measure by using tape at the axillary, xiphoid process, and umbrilical level

CONTACTS AND LOCATIONS:
Overall Officials: Saikaew Chuachan, Principal Investigator — Department of Physical Therapy, Faculty of Medicine, PSU; Natcha Kimthiaw, Bsc.PT, Study Director — Department of Physical Therapy, Faculty of Medicine, PSU; Luksamee Kaewchano, Bsc.PT, Study Director — Department of Physical Therapy, Faculty of Medicine, PSU; Ittiphon Pannarai, Bsc.PT, Study Director — Department of Physical Therapy, Faculty of Medicine, PSU; Jatuporn Jaturawanit, Bsc.PT, Study Director — Physical Therapy unit, Songklanakarind Hospital; Jitsupa Kittarakul, Bsc.PT, Study Director — Physical Therapy unit, Songklanakarind Hospital; Boonmas Chansirimongkol, B.N.S., Study Director — Medical Respiratory Care Unit, Prince of Songklanakarind Hospital; Kwankamol Kalsri, B.N.S, Study Director — Medical Respiratory Care Unit, Prince of Songklanakarind Hospital; Assoc.Prof.Siwasak Juthong, MD, Study Director — Division of Respiratory and Respiratory Critical Care Medicine, Department of Internal Medicine, PSU
Locations (1):
- Medical Respiratory Care Unit (MRCU), Prince of Songklanakarind Hospital, Songkhla, Thailand